CLINICAL TRIAL: NCT02027558
Title: Novel Treatment of Comorbid Insomnia and Sleep Apnea in Older Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 12-353
Record Dates: First submitted 2013-12-11; First posted 2014-01-06 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Insomnia; Apnea
Keywords: cognitive behavioral therapy; insomnia; apnea
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Apnea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral treatment (Experimental): Manual-based cognitive behavioral treatment focusing on sleep, sleep apnea, and PAP adherence provided by allied health personnel in individual sessions.
  Interventions: Behavioral: Insomnia treatment & PAP adherence
- Active control (Active Comparator): Manual-based non-directive general sleep education program provided by allied health personnel in individual sessions.
  Interventions: Behavioral: General sleep education

INTERVENTIONS:
Behavioral: Insomnia treatment & PAP adherence — Manual-based cognitive behavioral treatment focusing on sleep, sleep apnea, and PAP adherence provided by allied health personnel in individual sessions.
  Arms: Behavioral treatment
Behavioral: General sleep education — Manual-based non-directive general sleep education program provided by allied health personnel in individual sessions.
  Arms: Active control

SUMMARY:
The purpose of this study is to determine whether a novel intervention combining cognitive behavioral therapy for insomnia plus a positive airway pressure (PAP) behavioral adherence program provided by allied health personnel for older Veterans with obstructive sleep apnea and comorbid insomnia improves nighttime sleep and PAP adherence.

DETAILED DESCRIPTION:
Sleep disturbance is common in older adults and is associated with increased healthcare utilization, more depressive symptoms, and other adverse effects on health-related quality of life. Obstructive sleep apnea (OSA) is a disorder characterized by repetitive episodes of complete or partial upper airway obstruction occurring during sleep. OSA increases in prevalence with age, and is associated with increased risk of cardiovascular disease, decreased quality of life, and increased mortality. Insomnia also increases in prevalence with age, and is associated with numerous adverse outcomes, including cognitive decline, decreased quality of life, increased healthcare costs and increased mortality. The diagnostic criteria for insomnia include a decreased ability to fall asleep or stay asleep, frequent nighttime awakening or poor quality sleep that is associated with daytime impairment such as fatigue, impaired attention, or daytime sleepiness. Increasing evidence suggests that insomnia often coexists with OSA, particularly in older adults, and predicts worse outcomes of OSA. Both OSA and insomnia have a higher prevalence among Veterans, compared to the general population.

Little is known of the best approaches to manage the large number of patients with coexisting OSA and comorbid insomnia. Guidelines for best practice typically address these conditions separately, where positive airway pressure (PAP) is the standard for the treatment of OSA, and cognitive behavioral therapy for insomnia (CBT-I) is considered first-line treatment for chronic insomnia. CBT-I is particularly recommended for insomnia in older adults, where adverse effects of sleeping medications are most problematic. Early adherence to PAP therapy (i.e., within the first week of PAP therapy) is one of the strongest predictors of long-term PAP adherence. However, adherence rates to PAP therapy in patients with OSA are low. In addition, CBT-I has not been widely implemented for treatment of insomnia (in part due to limited access to mental health specialists able to provide CBT-I), untreated OSA limits response to treatment of insomnia, and untreated insomnia negatively impacts PAP adherence.

Based on this evidence and findings from the investigators' prior work, the investigators believe that an integrated, behavioral treatment approach which addresses both OSA and insomnia early in the course of PAP therapy is needed to maximize patient adherence and treatment success when these conditions coexist. The investigators propose a randomized controlled trial to test a novel, behavioral approach integrating best practices for management of both conditions among older Veterans with OSA who are prescribed PAP therapy and have comorbid insomnia. The purpose of this project is to determine whether this intervention improves nighttime sleep and PAP adherence.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for insomnia
* Diagnosis of obstructive sleep apnea (AHI > or = 15) and prescription of PAP therapy
* Age > or =50
* Community-dwelling
* Live within a 30-mile radius of VA GLAHS
* Have transportation to VA GLAHS to attend the intervention/control programs

Exclusion Criteria:

* Significant cognitive impairment (MMSE < 24)
* History of mania, major psychopathology or a psychiatric hospitalization in prior two years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Alessi, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (2):
- United States (2):
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fung CH, Martin JL, Josephson K, Fiorentino L, Dzierzewski JM, Jouldjian S, Tapia JC, Mitchell MN, Alessi C. Efficacy of Cognitive Behavioral Therapy for Insomnia in Older Adults With Occult Sleep-Disordered Breathing. Psychosom Med. 2016 Jun;78(5):629-39. doi: 10.1097/PSY.0000000000000314. PMID 27136498
- [Derived] Alessi CA, Fung CH, Dzierzewski JM, Fiorentino L, Stepnowsky C, Rodriguez Tapia JC, Song Y, Zeidler MR, Josephson K, Mitchell MN, Jouldjian S, Martin JL. Randomized controlled trial of an integrated approach to treating insomnia and improving the use of positive airway pressure therapy in veterans with comorbid insomnia disorder and obstructive sleep apnea. Sleep. 2021 Apr 9;44(4):zsaa235. doi: 10.1093/sleep/zsaa235. PMID 33221910

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Treatment | Active Control
Started | 62 | 63
Post-treatment | 49 | 60
3-month Follow-up | 53 | 58
6-month Follow-up | 53 | 61
Completed | 53 | 61
Not Completed | 9 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 4 | 1
Not completed — Refused assessment | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Behavioral Treatment: Manual-based cognitive behavioral treatment focusing on sleep, sleep apnea, and PAP adherence education program provided by allied health personnel in individual sessions.
- Total: Total of all reporting groups
Arm/Group | Behavioral Treatment | Active Control | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (6.7) | 63.7 (7.6) | 63.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 61 | 58 | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 17 | 31
  White | 35 | 34 | 69
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 4 | 2 | 6
Sleep quality [Mean (Standard Deviation); unit: units on a scale] — Total score on Pittsburgh Sleep Quality Index. Scores range from 0 to 21. Higher scores indicate worse outcome
  units on a scale | 11.0 (3.9) | 11.4 (4.4) | 11.2 (4.1)
Sleep onset latency from diary [Mean (Standard Deviation); unit: minutes] — Minimum value is 0 minutes. Maximum possible value is 1,440 minutes (24 hours). Higher scores indicate worse outcome.
  minutes | 40.9 (41.1) | 37.7 (27.3) | 39.3 (34.7)
Wake after sleep onset from sleep diary [Mean (Standard Deviation); unit: minutes] — Minimum value is 0 minutes. Maximum possible value is 1,440 minutes (24 hours). Higher scores indicate worse outcome.
  minutes | 53.4 (49.6) | 58.5 (58.7) | 56.0 (54.2)
Sleep efficiency from sleep diary [Mean (Standard Deviation); unit: percentage of time] — Sleep efficiency (mean percent time asleep while in bed) is calculated from 7 days of self-reported sleep diary. Higher percentages indicate better sleep outcome.
  percentage of time | 70.1 (17.8) | 69.9 (14.0) | 70.0 (15.9)
Sleep efficiency from wrist actigraphy [Mean (Standard Deviation); unit: percentage of time] — Sleep efficiency (mean percent time asleep while in bed) is calculated from 7 days of wrist actigraphy. Higher percentages indicate better sleep outcome.
  percentage of time | 77.7 (9.0) | 78.1 (10.9) | 77.9 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality
Description: Total score on the Pittsburgh Sleep Quality Index will be used as a measure of sleep quality. Scores range from 0 to 21. Higher scores indicate worse outcome.
Time Frame: Three months after randomization
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Behavioral Treatment: Manual-based cognitive behavioral treatment focusing on sleep, sleep apnea, and PAP adherence provided by allied health personnel in individual sessions.
  .
- Active Control: Manual-based non-directive general sleep education program provided by allied health personnel in individual sessions.
  .
Arm/Group | Behavioral Treatment | Active Control
Number analyzed (Participants) | 62 | 63
score on a scale | 6.25 (0.56) | 9.87 (0.53)
Statistical Analysis 1: Comparison: Behavioral Treatment vs Active Control; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Net) = -3.21, 95% CI 2-sided [-4.58 to -1.83], Standard Error of Mean 0.70 — The parameter estimate is the improvement in the outcome from baseline to 3-months for the treatment group versus the same improvement in respect to the control group

2. Primary Outcome: Sleep Onset Latency From Sleep Diary
Description: Sleep onset latency (minutes to fall asleep) will be calculated from 7 days of self-reported sleep diary. Minimum value is 0 minutes. Maximum possible value is 1,440 minutes (24 hours). Higher scores indicate worse outcome.
Time Frame: Three months after randomization
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Behavioral Treatment | Active Control
Number analyzed (Participants) | 62 | 63
minutes | 22.80 (3.86) | 35.77 (3.74)
Statistical Analysis 1: Comparison: Behavioral Treatment vs Active Control; Test type: Superiority; p = 0.013, Mixed Models Analysis; Mean Difference (Net) = -16.23, 95% CI 2-sided [-29.02 to -2.49], Standard Error of Mean 6.52 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Wake After Sleep Onset From Sleep Diary
Description: Wake after sleep onset (minutes awake from sleep onset to get up time) will be calculated from 7 days of self-reported sleep diary. Minimum value is 0 minutes. Maximum possible value is 1,440 minutes (24 hours). Higher scores indicate worse outcome.
Time Frame: Three months after randomization
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Behavioral Treatment | Active Control
Number analyzed (Participants) | 62 | 63
minutes | 20.42 (4.31) | 40.67 (4.16)
Statistical Analysis 1: Comparison: Behavioral Treatment vs Active Control; Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Net) = -20.46, 95% CI 2-sided [-37.63 to -3.29], Standard Error of Mean 8.75 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Sleep Efficiency From Sleep Diary
Description: Sleep efficiency (mean percent time asleep while in bed) will be calculated from 7 days of self-reported sleep diary. Scores range from 0 to 100 percent. Higher scores indicate better outcome.
Time Frame: Three months after randomization
Measure: Mean (Standard Error); unit: percentage of time
Arm/Group | Behavioral Treatment | Active Control
Number analyzed (Participants) | 62 | 63
percentage of time | 86.24 (1.69) | 75.69 (1.64)
Statistical Analysis 1: Comparison: Behavioral Treatment vs Active Control; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = 10.49, 95% CI 2-sided [4.53 to 16.44], Standard Error of Mean 3.04 — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Sleep Efficiency From Wrist Actigraphy
Description: Sleep efficiency (mean percent time asleep while in bed) will be calculated from 7 days of wrist actigraphy. Scores range from 0 to 100 percent. Higher scores indicate better outcome.
Time Frame: Three months after randomization
Measure: Mean (Standard Error); unit: percentage of time
Arm/Group | Behavioral Treatment | Active Control
Number analyzed (Participants) | 62 | 63
percentage of time | 81.70 (1.07) | 78.51 (1.07)
Statistical Analysis 1: Comparison: Behavioral Treatment vs Active Control; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = 4.35, 95% CI 2-sided [1.87 to 6.83], Standard Error of Mean 1.26 — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: PAP Adherence
Description: Number of nights positive airway pressure (PAP) was used >=4 hours during the first 90 days measured by remote monitoring. Scores range from 0 to 90 days. Higher scores indicate better outcome.
Time Frame: Three months after randomization
Measure: Mean (Standard Error); unit: number of nights
Arm/Group | Behavioral Treatment | Active Control
Number analyzed (Participants) | 62 | 63
number of nights | 38.58 (3.89) | 21.16 (3.14)
Statistical Analysis 1: Comparison: Behavioral Treatment vs Active Control; Test type: Superiority; p = 0.0007, t-test, 2 sided; Mean Difference (Final Values) = -17.42, 95% CI 2-sided [-27.29 to -7.55], Standard Error of Mean 4.99

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 6 months.
Arm/Group | Behavioral Treatment | Active Control
All-Cause Mortality (participants affected / at risk) | 0/62 | 1/63
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/63
Other Adverse Events (participants affected / at risk) | 1/62 | 0/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Treatment (N=62) | Active Control (N=63)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin irritation from wrist actigraph band.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT02027558/Prot_SAP_000.pdf